CLINICAL TRIAL: NCT07365540
Title: According to the WANFANG H Holistic Care Program - Clinical Training Group 113-WFHHCE-03 Program, Studies With a Start Date Before July 31, 2026, Are Eligible for the Relevant Criteria.。
Brief Title: The Effectiveness of Gamified Scenario-based Teaching in Improving Nurses' Awareness and Confidence in Clinical Emergency Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: N202504017; Holistic Care Program - Clinic (Other Grant/Funding Number: Holistic Care Program - Clinical Training Group 113-WFHHCE-03 program)
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamified Contextual Teaching (Experimental): The effectiveness of gamified scenario-based teaching in improving nurses' awareness and confidence in clinical emergency care
  Interventions: Other: gamified scenario-based teaching

INTERVENTIONS:
Other: gamified scenario-based teaching — A randomized controlled trial design was used, employing convenient sampling to recruit 68 nurses from a general ward of a medical center in northern Taiwan. Research tools included demographic and related data, an emergency knowledge scale, a self-confidence scale, and satisfaction assessment

SUMMARY:
Research Objective: This study aims to explore the effectiveness of gamified situational teaching in improving nurses' awareness and confidence in clinical emergency response.

ELIGIBILITY:
Convenience sampling was adopted, and the inclusion criteria included: nurses with more than 3 months of experience working in general wards; the exclusion criteria included: nurses in pediatric-related wards (including neonatal observation rooms and pediatric intensive care units).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
First Aid Skills Questionnaire | one month
  This study used a randomized controlled trial design. Blocked randomization was employed, dividing participants into an experimental group (gamified learning) and a control group (online video instruction). The experimental group learned first aid techniques using gamified learning, which involved taking photos of clinical first aid scenarios and placing them into the application. The application then transformed the photos into story scenarios, which the experimental group members would then immerse themselves in. The control group received instruction using existing online videos from the hospital.Two groups were enrolled using the hospital's emergency medical knowledge questionnaire at three stages: before intervention, after intervention, and one month after intervention. The questionnaire consisted of 10 multiple-choice questions. A correct answer was worth 10 points, while an incorrect answer or an answer that did not know was worth 0 points. The total score ranged from 0 to 100

SECONDARY OUTCOMES:
Confidence Scale | one month
  The C-scale (Grundy, 1993) was used for measurement. This scale has been translated into Chinese by scholars. The scale has a Cronbach's α value of 0.91 and a CVI value of 1.0, indicating good quantity-response reliability and validity. This scale consists of five items, with each item scored from one to five points, for a total score of 5 to 25 points. Higher scores indicate greater confidence in the research subjects' emergency treatment and techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Wanfang Hospital, Taipei, Taiwan